CLINICAL TRIAL: NCT03675659
Title: Effect of Magnesium Sulfate on Pain and Clicking Sound on Patients With Temporomandibular Joint Dysfunction
Brief Title: Intra-articular Magnesium Sulfate for Tmj Dysfunction
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Atef Fouda, prof of maxillofacial surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CD5618
Record Dates: First submitted 2018-09-15; First posted 2018-09-18 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Temporomandibular Joint Disorders; Temporomandibular Sprain
Keywords: tmj pain
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Injections, Intra-Articular; Prolotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intra-articular injection (Active Comparator): intra-articular injection with magnesium sulfate at weekly interval for four weeks
  Interventions: Drug: intra-articular injection
- control (Placebo Comparator): intra-articular injection with saline
  Interventions: Drug: intra-articular injection

INTERVENTIONS:
Drug: intra-articular injection — intra-articular injection with magnesium sulfate with four injections at weekly intervals
  Other Names: prolotherapy

SUMMARY:
mixing the magnesium sulfate with dextrose for management of tmj pain will be studied using intra-articular injection of the solution

ELIGIBILITY:
Inclusion Criteria:

* healthy females-no treatment received within the last 6 months-accept treatment protocol

Exclusion Criteria:

* unco-operative patients-patients with auto-immune diseases-patients diagnosed with arthritis

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females more affected than males
Enrollment: 100 (Estimated)
Dates: Start 2017-09-09 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
estimation of pain: Visual Analog Scale | one year
  Visual Analog Scale pain measurement with "0" indicates no pain and "100" the maximum pain felt ever

CONTACTS AND LOCATIONS:
Locations (1):
- Atef, Giza, Egypt